CLINICAL TRIAL: NCT07043725
Title: A Randomized, Open-label, Multicenter, Parallel-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of TQB2102 for Injection Versus TCbHP in Neoadjuvant Treatment of Breast Cancer With Positive HER2 Expression
Brief Title: A Clinical Study of Neoadjuvant Treatment With TQB2102 for Injection for Human Epidermal Growth Factor Receptor 2 (HER2) Positive Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-III-05
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Injections; Trastuzumab; pertuzumab; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2102 for injection (Experimental): 6mg/kg TQB2102 for injection, Intravenous infusion, administered every 3 weeks, 21 days as a treatment cycle, 8 cycles.
  Interventions: Drug: TQB2102 for injection
- Trastuzumab injection and Pertuzumab Injection and Docetaxel Injection and Carboplatin Injection (Active Comparator): Trastuzumab injection (The first dose is 8mg/kg, followed by 6mg/kg), Pertuzumab Injection (The first dose is 840, followed by 420mg), Docetaxel Injection (75mg/m2 ) combined with Carboplatin Injection (AUC-6, 800 mg max), Intravenous infusion, administered every 3 weeks, 21 days as a treatment cycle, 6 cycles.
  Interventions: Drug: Trastuzumab injection and Pertuzumab Injection and Docetaxel Injection and Carboplatin Injection

INTERVENTIONS:
Drug: TQB2102 for injection — TQB2102 for injection is a HER2 dual-antibody-drug Conjugate (ADC)
  Arms: TQB2102 for injection
Drug: Trastuzumab injection and Pertuzumab Injection and Docetaxel Injection and Carboplatin Injection — TCbHP is a commonly used chemotherapy scheme for HER2 positive breast cancer. H represents Trastuzumab injection, P represents Pertuzumab Injection, T represents Docetaxel injection and C represents Carboplatin injection.
  Arms: Trastuzumab injection and Pertuzumab Injection and Docetaxel Injection and Carboplatin Injection

SUMMARY:
This is a randomized, open, positive drug control, multi center phase III study. Through the evaluation of tpCR, bpCR, ORR, EFS, IDFS, OS , AEs and other indicators, it proves the effectiveness and safety of TQB2102 for injection versus TCbHP in the neoadjuvant treatment of HER2 positive breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this study, sign the informed consent form, and have good compliance;
* Eastern Cooperative Oncology Group performance status (ECOG PS) score: 0-1; expected survival >6 months;
* Histologically or cytologically confirmed HER2-positive invasive breast cancer;
* Hormone receptor (HR) status confirmed;
* Clinical stage at diagnosis: T2-4 with any N, M0, or any T with N1-3, M0;
* Agree to undergo breast cancer resection if meeting surgical criteria after neoadjuvant therapy;
* Major organ function is adequate, meeting specific criteria;
* Must agree to use contraception during the study and for 6 months after study completion; female patients must have a negative serum pregnancy test within 7 days before enrollment and must not be lactating; male subjects must agree to use contraception during the study and for 6 months after study completion

Exclusion Criteria:

* Stage IV metastatic breast cancer or other cases judged by the investigator as unsuitable for radical surgical resection after neoadjuvant therapy;
* Bilateral breast cancer or inflammatory breast cancer;
* History of invasive breast cancer or ductal carcinoma in situ;
* Prior anti-tumor therapy for breast cancer, including chemotherapy, endocrine therapy, targeted therapy, radiotherapy, surgery, etc.;
* Comorbidities and medical history:

  * Other malignancies within 5 years or currently;
  * Adverse reactions from prior treatment not recovered to CTCAE v5.0 grade ≤1;
  * Major surgery, significant traumatic injury within 4 weeks before first dose, or anticipated major surgery during the study, or unhealed wounds/fractures;
  * Conditions affecting intravenous injection or blood sampling;
  * Congenital bleeding or coagulation disorders, or bleeding/coagulation disorders within 28 days before study treatment, or use of aspirin >325 mg/day (maximum antiplatelet dose), dipyridamole, ticlopidine, clopidogrel, or cilostazol within 7 days before study treatment;
  * Arterial/deep venous thrombotic events within 6 months before first dose, e.g., cerebrovascular accident, deep vein thrombosis, pulmonary embolism;
  * Poorly controlled blood pressure (systolic ≥150 mmHg or diastolic ≥100 mmHg);
  * Significant cardiovascular disease, including；
  * Uncontrolled ≥CTCAE grade 2 infection within 14 days before study treatment;
  * History of interstitial lung disease/pneumonitis (non-infectious) requiring steroid treatment, current interstitial lung disease/pneumonitis, or suspected interstitial lung disease/pneumonitis on screening imaging that cannot be ruled out;
* Tumor-related symptoms and treatment:

  * Prior excisional biopsy of primary tumor and/or axillary lymph nodes or sentinel lymph node biopsy before study treatment;
  * Surgery, chemotherapy, radiotherapy, or other anti-tumor therapy within 3 weeks before study treatment (washout period calculated from last treatment);
  * Prior taxane or carboplatin therapy for any malignancy;
  * Treatment with National Medical Products Administration-approved traditional Chinese medicine with clear anti-tumor indications within 2 weeks before study treatment.
* Study treatment-related:

  * Severe hypersensitivity to monoclonal antibodies;
  * Uncontrolled active autoimmune disease within 2 weeks before study treatment;
  * Allergy to any study drug or its components/excipients;
  * Live vaccination within 28 days before study treatment, including measles, mumps, rubella, varicella, yellow fever, seasonal flu, Influenza A virus subtype (H1N1) flu, rabies, Bacille Calmette-Guerin vaccine (BCG), and typhoid vaccines.
* Any condition judged by the investigator to jeopardize subject safety or study completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Rate of total physiological complete response (tpCR) evaluated by Independent Review Committee (IRC) | Up to 26 months after study start
  Rate of subjects with no residual invasive cancer in the primary breast lesion and negative regional lymph nodes upon microscopic examination after primary tumor resection, as assessed by IRC.

SECONDARY OUTCOMES:
Rate of total physiological complete response (tpCR) evaluated by the investigator | Up to 24 months after study start
  Rate of subjects with no residual invasive cancer in the primary breast lesion and negative regional lymph nodes upon microscopic examination after primary tumor resection, as assessed by the investigator.
Breast pathological complete response (bpCR) evaluated by IRC and the investigator | Up to 26 months after study start
  Percentage of subjects with no residual invasive cancer in the primary breast lesion upon microscopic examination after primary tumor resection, as assessed by IRC and the investigator.
Objective response rate (ORR) | Up to 22 months after study start
  The percentage of subjects achieving complete response (CR) or partial response (PR) as assessed by the investigator based on the Response Evaluation Criteria In Solid Tumors (RECIST 1.1) .
There year Event-free survival (EFS) | Up to 50 months after study start
  Time from randomization to the first occurrence of any of the following events: ipsilateral or contralateral invasive breast cancer recurrence, regional or distant invasive breast cancer recurrence, or death from any cause.
There year Invasive Disease-free survival (IDFS) | Up to 50 months after study start
  Time from randomization to the first occurrence of any of the following events: ipsilateral or contralateral invasive breast cancer recurrence, regional or distant invasive breast cancer recurrence, or death from any cause.
Overall Survival (OS) | Up to 50 months after study start
  Time from randomization to death due to any cause.
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and indicators of abnormal laboratory tests | From the date of signing the informed consent to 40 days after the last dosing or radical mastectomy for breast cancer or a new anti-tumor treatment, whichever comes first.
  To evaluate the safety of TQB2102 for Injection compared to TCbHP in the neoadjuvant treatment of HER2 positive early breast cancer, including: the incidence and severity of adverse events (AEs), abnormal laboratory test values, and serious adverse events (SAEs).
Incidence of Anti-drug antibody (ADA) and neutralizing antibodies (NAb) | Up to 22 months after study start
  Incidence of ADA and Nab

CONTACTS AND LOCATIONS:
Locations (76):
- China (76):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical University, Wuhu, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Cancer Hospital Affiliated to Chongqing University, Chongqing Cancer Hospital, Chongqing Cancer Research Institute, and Chongqing Cancer Center, Chongqing, Chongqing Municipality
  - The First Hospital Affiliated to Army Medical University, Chongqing, Chongqing Municipality
  - Quanzhou First Hospital, Quanzhou, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Zhongshan Hospital Xiamen university, Xiamen, Fujian
  - ZhangZhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Gansu Provincial Academic Institute for Medical Research, Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - Guigang City People's Hospital, Guigang, Guangxi
  - Guangxi Cancer Institutu (Guangxi Cancer Hospital, Guangxi Medical University Cancer Hospital, Guangxi Cancer Center), Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - First Hospital of QinHuangDao, Qinhuangdao, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Jiamusi Cancer Hospital, Jiamusi, Heilongjiang
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjinag
  - Anyang Tumor Hospital, Anyang, Henan
  - The People's Hospital of Anyang City, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Xiangya Hospital ZhuZhou Central South University, Zhuzhou, Hunan
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - NanChang People's Hospital, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of the Air Force Medical University of the People's Liberation Army, Xi'an, Shaanxi
  - The Second Affiliated Hospital of the Air Force Medical University of the People's Liberation Army, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Cancer Hospital of Shandong First Medical University, Shandong Cancer Institute, Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Taian, Shandong
  - WeiFang People's Hospital, Weifang, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - The Second People's Hospital of YiBin, Yibin, Sichuan
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Medical University Cancer Hospital, Ürümqi, Xinjiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang